CLINICAL TRIAL: NCT02335424
Title: A Phase II Clinical Trial of Pembrolizumab (MK-3475) in Subjects With Advanced/Unresectable or Metastatic Urothelial Cancer
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Advanced Urothelial Cancer (MK-3475-052/KEYNOTE-052)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-052; MK-3475-052 (Other: Merck Protocol Number); KEYNOTE-052 (Other: Merck); 2014-002206-20 (EudraCT Number)
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Urothelial Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); bladder cancer
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body; Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 2 years. Eligible participants who stopped the initial course of pembrolizumab due to complete response (CR) or completed initial course of pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to an additional year.
  Interventions: Biological: pembrolizumab

INTERVENTIONS:
Biological: pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
This is a study using pembrolizumab (MK-3475, KEYTRUDA®) for first-line treatment of participants with advanced/unresectable (inoperable) or metastatic urothelial cancer who are ineligible for cisplatin-based therapy. The primary study objective is to determine the objective response rate (ORR) in all participants and by programmed cell death ligand 1 (PD-L1) status.

With Amendment 4, once a participant has achieved the study objective or the study has ended, the participant will be discontinued from this study and will be enrolled in an extension study to continue protocol-defined assessments and treatment.

DETAILED DESCRIPTION:
Participants receiving pembrolizumab who attain a complete response (CR) may consider stopping trial treatment if they meet criteria for holding therapy. Participants who stop trial treatment after receiving 24 months of trial treatment for reasons other than progressive disease (PD) or intolerability, or participants who attain a CR and stop trial treatment may be eligible for up to one year of retreatment upon experiencing PD.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of advanced/unresectable (inoperable) or metastatic urothelial cancer of the renal pelvis, ureter, bladder, or urethra (transitional cell and mixed transitional/non-transitional cell histologies)
* Ineligible for cisplatin therapy
* No prior systemic chemotherapy for metastatic disease (adjuvant or neoadjuvant platinum-based chemotherapy with recurrence >12 months since completion of therapy is allowed)
* Available tissue from a newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Adequate organ function
* Female participants of childbearing potential have a negative urine or serum pregnancy test; surgically sterile, or willing to use 2 acceptable methods of birth control, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study treatment
* Male participants must be willing to use an adequate method of contraception starting with the first dose of study medication through 120 days after the last dose of study treatment

Exclusion Criteria:

* Disease that is suitable for local therapy administered with curative intent
* Currently participating or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of study treatment
* Prior anti-cancer monoclonal antibody (mAb) for direct anti-neoplastic treatment within 4 weeks prior to study Day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or not recovered from AEs due to a previously administered agent
* Known additional malignancy that is progressing or requires active treatment excepting basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in past 2 years
* Evidence of interstitial lung disease or active non-infectious pneumonitis
* Active infection requiring systemic therapy
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of study treatment
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another co-inhibitory T-cell receptor
* Known human immunodeficiency virus (HIV)
* Known active Hepatitis B or C
* Received a live virus vaccine within 30 days of planned start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Balar AV, Castellano D, O'Donnell PH, Grivas P, Vuky J, Powles T, Plimack ER, Hahn NM, de Wit R, Pang L, Savage MJ, Perini RF, Keefe SM, Bajorin D, Bellmunt J. First-line pembrolizumab in cisplatin-ineligible patients with locally advanced and unresectable or metastatic urothelial cancer (KEYNOTE-052): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2017 Nov;18(11):1483-1492. doi: 10.1016/S1470-2045(17)30616-2. Epub 2017 Sep 26. PMID 28967485
- [Result] Vuky J, Balar AV, Castellano D, O'Donnell PH, Grivas P, Bellmunt J, Powles T, Bajorin D, Hahn NM, Savage MJ, Fang X, Godwin JL, Frenkl TL, Homet Moreno B, de Wit R, Plimack ER. Long-Term Outcomes in KEYNOTE-052: Phase II Study Investigating First-Line Pembrolizumab in Cisplatin-Ineligible Patients With Locally Advanced or Metastatic Urothelial Cancer. J Clin Oncol. 2020 Aug 10;38(23):2658-2666. doi: 10.1200/JCO.19.01213. Epub 2020 Jun 17. PMID 32552471
- [Derived] Topp BG, Channavazzala M, Mayawala K, De Alwis DP, Rubin E, Snyder A, Wolchok JD, Ribas A. Tumor dynamics in patients with solid tumors treated with pembrolizumab beyond disease progression. Cancer Cell. 2023 Sep 11;41(9):1680-1688.e2. doi: 10.1016/j.ccell.2023.08.004. PMID 37699333
- [Derived] Balar AV, Castellano DE, Grivas P, Vaughn DJ, Powles T, Vuky J, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Necchi A, Petrylak DP, Plimack ER, Xu JZ, Imai K, Moreno BH, Bellmunt J, de Wit R, O'Donnell PH. Efficacy and safety of pembrolizumab in metastatic urothelial carcinoma: results from KEYNOTE-045 and KEYNOTE-052 after up to 5 years of follow-up. Ann Oncol. 2023 Mar;34(3):289-299. doi: 10.1016/j.annonc.2022.11.012. Epub 2022 Dec 6. PMID 36494006
- [Derived] Bellmunt J, de Wit R, Fradet Y, Climent MA, Petrylak DP, Lee JL, Fong L, Necchi A, Sternberg CN, O'Donnell PH, Powles T, Plimack ER, Bajorin DF, Balar AV, Castellano D, Choueiri TK, Culine S, Gerritsen W, Gurney H, Quinn DI, Vuky J, Vogelzang NJ, Cristescu R, Lunceford J, Saadatpour A, Loboda A, Ma J, Rajasagi M, Godwin JL, Homet Moreno B, Grivas P. Putative Biomarkers of Clinical Benefit With Pembrolizumab in Advanced Urothelial Cancer: Results from the KEYNOTE-045 and KEYNOTE-052 Landmark Trials. Clin Cancer Res. 2022 May 13;28(10):2050-2060. doi: 10.1158/1078-0432.CCR-21-3089. PMID 35247908
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible to receive second course treatment with pembrolizumab if they met criteria for re-treatment. Per protocol, only data generated during the initial course of treatment contributed to efficacy and safety outcome measures.
Pre-assignment Details: Results are based on a database cutoff date of 18-February-2022.
Groups:
- Pembrolizumab 200 mg: Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to 2 years. Eligible participants who stopped the initial course of pembrolizumab due to complete response (CR) or completed initial course of pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to an additional year.
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg
Started | 374
Treated | 370
Received Second Course Treatment | 13
Completed | 0
Not Completed | 374
Not completed — Withdrawal by Subject | 19
Not completed — Adverse Event | 25
Not completed — Death | 273
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 13
Not completed — Participation in study terminated by Sponsor | 39
Not completed — Protocol Violation | 1
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all allocated participants.
Groups:
- Pembrolizumab 200 mg: Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 2 years. Eligible participants who stopped the initial course of pembrolizumab due to complete response (CR) or completed initial course of pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to an additional year.
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 374
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 326
  Unknown or Not Reported | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 332
  More than one race | 2
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: ORR was determined in all participants and was defined as the percentage of participants who had a confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). Participants with missing data were considered non-responders. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Percentage of participants | 28.9 [24.3 to 33.8]

2. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1%
Description: ORR was determined in participants who had a PD-L1 CPS of ≥1% as measured by immunohistochemistry assay. ORR was defined as the percentage of participants who had a confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). Participants with missing data were considered non-responders. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment, during the initial course of treatment, and had a PD-L1 positive expression of ≥1% CPS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 282
Percentage of participants | 32.6 [27.2 to 38.4]

3. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥10%
Description: ORR was determined in participants who had a PD-L1 CPS of ≥10% as measured by immunohistochemistry assay. ORR was defined as the percentage of participants who had a confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). Participants with missing data were considered non-responders. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment, during the initial course of treatment, and had a PD-L1 strong positive expression of ≥10% CPS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 110
Percentage of participants | 47.3 [37.7 to 57.0]

4. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: DOR was determined in participants who demonstrated a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death and was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants who had not progressed or died at the time of analysis were censored at the date of their last tumor assessment. Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment, during the initial course of treatment, and who had a confirmed CR or confirmed PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 107
Months | 33.4 [18.2 to 48.7]

5. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1%
Description: DOR was determined in participants who had a PD-L1 CPS of ≥1%, as measured by immunohistochemistry assay, and had a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death and was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants who had not progressed or died at the time of analysis were censored at the date of their last tumor assessment. Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment during the initial course of treatment, had a PD-L1 positive expression of ≥1% CPS, and who had a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 92
Months | 35.8 [20.4 to NA] — NA = upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse

6. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥10%
Description: DOR was determined in participants who had a PD-L1 CPS of ≥10%, as measured by immunohistochemistry assay, and had a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). DOR was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death and was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants who had not progressed or died at the time of analysis were censored at the date of their last tumor assessment. Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment during the initial course of treatment, had a PD-L1 strong positive expression of ≥10% CPS, and who had a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 52
Months | NA [18.1 to NA] — NA = median and upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse

7. Secondary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: PFS was determined in all participants. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Time to scheduled tumor assessment visit rather than the actual tumor assessment visit was used in the analysis. PFS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment during the initial course of treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Months | 2.5 [2.1 to 3.4]

8. Secondary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1%
Description: PFS was determined in participants who had a PD-L1 CPS of ≥1% as measured by immunohistochemistry assay. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Time to scheduled tumor assessment visit rather than the actual tumor assessment visit was used in the analysis. PFS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 282
Months | 3.4 [2.3 to 4.0]

9. Secondary Outcome: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥10%
Description: PFS was determined in participants who had a PD-L1 CPS of ≥10% as measured by immunohistochemistry assay. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per RECIST 1.1 as assessed by Blinded Independent Central Review (BICR). Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Time to scheduled tumor assessment visit rather than the actual tumor assessment visit was used in the analysis. PFS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 110
Months | 4.9 [3.8 to 10.8]

10. Secondary Outcome: Overall Survival (OS) in All Participants
Description: OS was determined for all participants and was defined as the time from randomization to death due to any cause. OS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Months | 11.3 [9.7 to 13.1]

11. Secondary Outcome: Overall Survival (OS) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1%
Description: OS was determined in participants who had a PD-L1 CPS of ≥1%, as measured by immunohistochemistry assay. OS was defined as the time from randomization to death due to any cause. OS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 282
Months | 12.4 [10.8 to 15.0]

12. Secondary Outcome: Overall Survival (OS) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥10%
Description: OS was determined in participants who had a PD-L1 CPS of ≥10% as measured by immunohistochemistry assay. OS was defined as the time from randomization to death due to any cause. OS was calculated using the product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 110
Months | 18.5 [12.2 to 28.5]

13. Secondary Outcome: Progression Free Survival Rate (PFS Rate) at Month 6 in All Participants
Description: The PFS rate was determined in all participants at Month 6. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR). Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Time to scheduled tumor assessment visit rather than the actual tumor assessment visit was used in the analysis. PFS at Month 6 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 6
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Percentage of participants | 34.0 [29.2 to 38.8]

14. Secondary Outcome: Progression Free Survival Rate (PFS Rate) at Month 6 in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1%
Description: The PFS rate was determined in participants who had a PD-L1 CPS of ≥1%, as measured by immunohistochemistry assay, at Month 6. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR). Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Time to scheduled tumor assessment visit rather than the actual tumor assessment visit was used in the analysis. PFS at Month 6 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 282
Percentage of participants | 37.9 [32.2 to 43.5]

15. Secondary Outcome: Progression Free Survival Rate (PFS Rate) at Month 6 in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥10%
Description: The PFS rate was determined in participants who had a PD-L1 CPS of ≥10%, as measured by immunohistochemistry assay, at Month 6. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR). Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Time to scheduled tumor assessment visit rather than the actual tumor assessment visit was used in the analysis. PFS at Month 6 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 110
Percentage of participants | 49.0 [39.4 to 57.9]

16. Secondary Outcome: Progression Free Survival Rate (PFS Rate) at Month 12 in All Participants
Description: The PFS rate was determined in all participants at Month 12. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR). Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Time to scheduled tumor assessment visit rather than the actual tumor assessment visit was used in the analysis. PFS at Month 12 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 12
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Percentage of participants | 22.9 [18.7 to 27.3]

17. Secondary Outcome: Progression Free Survival Rate (PFS Rate) at Month 12 in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1%
Description: The PFS rate was determined in participants who had a PD-L1 CPS of ≥1%, as measured by immunohistochemistry assay, at Month 12. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR). Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Time to scheduled tumor assessment visit rather than the actual tumor assessment visit was used in the analysis. PFS at Month 12 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 282
Percentage of participants | 25.8 [20.8 to 31.1]

18. Secondary Outcome: Progression Free Survival Rate (PFS Rate) at Month 12 in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥10%
Description: The PFS rate was determined in participants who had a PD-L1 CPS of ≥10%, as measured by immunohistochemistry assay, at Month 12. PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR). Per RECIST 1.1, PD was a ≥20% increase in the sum of diameters of target lesions plus an absolute increase of ≥5 mm in the sum, or the appearance of ≥1 new lesions. Time to scheduled tumor assessment visit rather than the actual tumor assessment visit was used in the analysis. PFS at Month 12 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 110
Percentage of participants | 38.6 [29.5 to 47.7]

19. Secondary Outcome: Overall Survival Rate (OS Rate) at Month 6 in All Participants
Description: The OS rate was determined for all participants at Month 6 and was defined as the time from randomization to death due to any cause. OS at Month 6 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 6
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Percentage of participants | 67.0 [62.0 to 71.5]

20. Secondary Outcome: Overall Survival Rate (OS Rate) at Month 6 in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1%
Description: The OS rate was determined in participants who had a PD-L1 CPS of ≥1%, as measured by immunohistochemistry assay, at Month 6. OS was defined as the time from randomization to death due to any cause. OS at Month 6 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 282
Percentage of participants | 71.3 [65.6 to 76.2]

21. Secondary Outcome: Overall Survival Rate (OS Rate) at Month 6 in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥10%
Description: The OS rate was determined in participants who had a PD-L1 CPS of ≥10%, as measured by immunohistochemistry assay, at Month 6. OS was defined as the time from randomization to death due to any cause. OS at Month 6 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 110
Percentage of participants | 76.3 [67.2 to 83.2]

22. Secondary Outcome: Overall Survival Rate (OS Rate) at Month 12 in All Participants
Description: The OS rate was determined for all participants at Month 12 and was defined as the time from randomization to death due to any cause. OS at Month 12 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 12
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Percentage of participants | 46.9 [41.8 to 51.9]

23. Secondary Outcome: Overall Survival Rate (OS Rate) at Month 12 in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1%
Description: The OS rate was determined in participants who had a PD-L1 CPS of ≥1%, as measured by immunohistochemistry assay, at Month 12. OS was defined as the time from randomization to death due to any cause. OS at Month 12 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 282
Percentage of participants | 50.9 [45.0 to 56.6]

24. Secondary Outcome: Overall Survival Rate (OS Rate) at Month 12 in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥10%
Description: The OS rate was determined in participants who had a PD-L1 CPS of ≥10%, as measured by immunohistochemistry assay, at Month 12. OS was defined as the time from randomization to death due to any cause. OS at Month 12 was calculated using product-limit (Kaplan-Meier) method for censored data. Participants were censored at the date of their last assessment. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Month 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 110
Percentage of participants | 60.7 [50.9 to 69.1]

25. Secondary Outcome: Programmed Cell Death Ligand 1 (PD-L1) Expression Status
Description: PD-L1 expression status was determined as the percent of disease tumor cells, from newly obtained tumor biopsies, demonstrating plasma membrane PD-L1 staining of any intensity using an immunohistochemistry (IHC) assay. The assay uses a Combined Positive Score (CPS) as a measure of PD-L1 positivity. The CPS is calculated as the number of PD-L1-positive cells divided by the number of viable tumor cells analyzed multiplied by 100. A CPS of <1% = negative; ≥1% = positive; and ≥10% = strongly positive. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Day 1
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Participants
  PD-L1 CPS <1% | 79
  PD-L1 CPS ≥1% to <10% | 172
  PD-L1 CPS ≥10% | 110
  Unknown | 9

26. Secondary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Participants | 361

27. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: as for outcome 26
Time Frame: Up to approximately 26 months
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Participants | 62

28. Other Pre Specified Outcome: Objective Response Rate (ORR) Per Modified Response Evaluation Criteria in Solid Tumors (Modified RECIST) in All Participants
Description: ORR was determined in all participants and was defined as the percentage of participants who had a confirmed Complete Response (CR: complete disappearance of all lesions and no new lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per modified RECIST as assessed by Blinded Independent Central Review (BICR). Modified RECIST differs from RECIST 1.1 in that progressive disease requires confirmation by a repeat radiological assessment no less than 4 weeks from the date of first documented progressive disease. Participants with missing data were considered non-responders. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment during the initial course of treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 370
Percentage of participants | 30.5 [25.9 to 35.5]

29. Other Pre Specified Outcome: Objective Response Rate (ORR) Per Modified Response Evaluation Criteria in Solid Tumors (Modified RECIST) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥1%
Description: ORR was determined in participants who had a PD-L1 CPS of ≥1% as measured by immunohistochemistry assay. ORR was defined as the percentage of participants who had a confirmed Complete Response (CR: complete disappearance of all lesions and no new lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per modified RECIST as assessed by Blinded Independent Central Review (BICR). Modified RECIST differs from RECIST 1.1 in that progressive disease requires confirmation by a repeat radiological assessment no less than 4 weeks from the date of first documented progressive disease. Participants with missing data were considered non-responders. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 282
Percentage of participants | 34.4 [28.9 to 40.3]

30. Other Pre Specified Outcome: Objective Response Rate (ORR) Per Modified Response Evaluation Criteria in Solid Tumors (Modified RECIST) in Participants With a Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) of ≥10%
Description: ORR was determined in participants who had a PD-L1 CPS of ≥10% as measured by immunohistochemistry assay. ORR was defined as the percentage of participants who had a confirmed Complete Response (CR: complete disappearance of all lesions and no new lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per modified RECIST as assessed by Blinded Independent Central Review (BICR). Modified RECIST differs from RECIST 1.1 in that progressive disease requires confirmation by a repeat radiological assessment no less than 4 weeks from the date of first documented progressive disease. Participants with missing data were considered non-responders. Per protocol, only data generated during the initial course of treatment contributed to the analysis.
Time Frame: Up to approximately 80.5 months
Population: All participants who received at least one dose of study treatment, during the initial course of treatment, and had a PD-L1 positive expression of ≥10% CPS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg
Number analyzed (Participants) | 110
Percentage of participants | 49.1 [39.4 to 58.8]

ADVERSE EVENTS:
Time Frame: Up to approximately 80.5 months
Description: Adverse events=all participants who received ≥1 dose of study treatment; all-cause mortality=all allocated participants. Per protocol, progression of cancer under study was not considered an AE unless related to study drug. MedDRA preferred terms "Neoplasm progression (NP)", "Malignant NP" & "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Second Course Pembrolizumab: Participants who met the criteria for retreatment received pembrolizumab 200 mg by IV infusion on Day 1 of each 21-day cycle for up to 1 year of treatment.
Arm/Group | Pembrolizumab | Second Course Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 305/374 | 8/13
Serious Adverse Events (participants affected / at risk) | 190/370 | 6/13
Other Adverse Events (participants affected / at risk) | 342/370 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=370) | Second Course Pembrolizumab (N=13)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Addison's disease (Endocrine disorders) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 5 (5) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Cardiac complication associated with device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 15 (15) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 9 (9) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 26 (31) | 0 (0)
Urosepsis (Infections and infestations) | 14 (14) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 13 (14) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 12 (13) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 5 (5) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 5 (5) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=370) | Second Course Pembrolizumab (N=13)
Anaemia (Blood and lymphatic system disorders) | 73 (84) | 3 (3)
Ear swelling (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 42 (42) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 47 (57) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 6 (6) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 87 (100) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 82 (121) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 23 (23) | 0 (0)
Nausea (Gastrointestinal disorders) | 77 (89) | 1 (1)
Vomiting (Gastrointestinal disorders) | 56 (79) | 0 (0)
Asthenia (General disorders) | 44 (49) | 0 (0)
Chest pain (General disorders) | 20 (22) | 0 (0)
Chills (General disorders) | 27 (31) | 0 (0)
Fatigue (General disorders) | 129 (156) | 0 (0)
Influenza like illness (General disorders) | 19 (21) | 0 (0)
Oedema (General disorders) | 6 (6) | 1 (1)
Oedema peripheral (General disorders) | 63 (74) | 1 (1)
Peripheral swelling (General disorders) | 7 (7) | 1 (1)
Pyrexia (General disorders) | 51 (64) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 16 (17) | 1 (1)
Tooth infection (Infections and infestations) | 2 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 19 (23) | 0 (0)
Urinary tract infection (Infections and infestations) | 76 (98) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 22 (26) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 27 (31) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 27 (31) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 27 (30) | 0 (0)
Blood creatinine increased (Investigations) | 53 (67) | 0 (0)
Inspiratory capacity decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 44 (47) | 2 (2)
White blood cell count decreased (Investigations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 102 (116) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 19 (19) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 37 (51) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 24 (29) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 (26) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (20) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 41 (53) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 (74) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 47 (55) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 26 (29) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (22) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 (31) | 0 (0)
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 35 (41) | 2 (2)
Headache (Nervous system disorders) | 20 (23) | 1 (1)
Insomnia (Psychiatric disorders) | 29 (29) | 0 (0)
Haematuria (Renal and urinary disorders) | 53 (63) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 16 (16) | 1 (1)
Proteinuria (Renal and urinary disorders) | 21 (23) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 76 (92) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 (57) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 87 (114) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 59 (83) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 20 (21) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT02335424/Prot_SAP_001.pdf